CLINICAL TRIAL: NCT02858037
Title: A Phase 3B Open-Label Follow-on Trial to Assess the Continued Safety of and Adherence to a Vaginal Ring Containing Dapivirine in Women
Brief Title: Trial to Assess the Continued Safety of and Adherence to a Vaginal Ring Containing Dapivirine in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTN-025
Record Dates: First submitted 2016-07-18; First posted 2016-08-08 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will receive a silicone elastomer vaginal matrix ring containing 25 mg of dapivirine to be replaced each month for a total period of 12 months of use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIV Open-label Prevention (Experimental): Following demonstration of safety and efficacy of the dapivirine vaginal ring in MTN-020, eligible MTN-020 participants will be offered enrollment into MTN-025, a trial designed to obtain additional safety and adherence data in women
  MTN-020:NCT01617096 MTN-025: NCT02858037
  Interventions: Combination Product: Dapivirine Vaginal Ring

INTERVENTIONS:
Combination Product: Dapivirine Vaginal Ring — Dapivirine Vaginal Ring, 25 ring given monthly for at least one year.

SUMMARY:
HIV Open-label Prevention Extension (HOPE).

DETAILED DESCRIPTION:
A Phase 3B Open-Label Follow-on Trial to Assess the Continues Safety of and Adherence to a Vaginal ring Containing Dapivirine in Women

ELIGIBILITY:
Inclusion Criteria:

Women must meet all of the following criteria to be eligible for inclusion in the study

1. Previously enrolled in MTN-020 (ASPIRE)
2. Able and willing to provide written informed consent to be screened for and to take part in the study
3. Able and willing to provide adequate locator information, as defined in site SOPs
4. HIV-uninfected based on testing performed by study staff at Screening and Enrollment
5. Using an effective method of contraception at Enrollment, and intending to use an effective method for the duration of study participation; effective methods include hormonal methods (except contraceptive ring); intrauterine contraceptive device (IUCD); and sterilization (of participant, as defined in site SOPs)
6. At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation

Exclusion Criteria:

Women who meet any of the following criteria will be excluded from the study

1. Study product use permanently discontinued in response to an AE or safety related concern while taking part in the MTN-020 (ASPIRE) trial
2. Per participant report at Screening:

   1. Plans to relocate away from the study site during study participation
   2. Plans to travel away from the study site for more than three consecutive months during study participation
3. Per participant report at Enrollment, currently taking Post-Exposure Prophylaxis (PEP)
4. With the exception of MTN-020 (ASPIRE), participation in any other research study involving drugs, medical devices, vaginal products, or vaccines, within 60 days of enrollment
5. Is pregnant at Screening/Enrollment or planning to become pregnant in the participant's anticipated study participation period
6. Currently breastfeeding
7. Diagnosed with urinary tract infection (UTI), pelvic inflammatory disease (PID), STI or reproductive tract infection (RTI) requiring treatment per WHO guidelines
8. At Screening, has a clinically apparent Grade 3 pelvic exam finding (observed by study staff) as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009), Addendum 1-Female Genital Grading Table for Use in Microbicide Studies
9. Has any of the following laboratory abnormalities at Screening Visit:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT) > Grade 3*
   2. Creatinine > Grade 3*
   3. Hemoglobin > Grade 3*
   4. Platelet count > Grade 3*
   5. Pap result ≥ Grade 3 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009)
10. Has any significant medical condition or other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

    -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1456 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Steytler, Study Director — International Partnership for Microbicides
Locations (17):
- Malawi (2):
  - Johns Hopkins University Research Project, Blantyre
  - Malawi Clinical Research Center, Lilongwe
- South Africa (10):
  - Medical Research Council of South Africa, Westville, Durban
  - WRHI Clinical Research Center, Johannesburg, Gauteng
  - Verulam Clinical Research Center, Durban, KwaZulu-Natal
  - Botha's Hill Clinical Research Center, Durban, KwaZulu-Natal
  - Chatsworth Clinical Research Center, Durban, KwaZulu-Natal
  - Isipingo Clinical Research Center, Durban, KwaZulu-Natal
  - Tongaat Clinical Research Center, Durban, KwaZulu-Natal
  - Emavundleni Research Centre, Cape Town, Western Cape
  - eThekwini Clinical Research Center, Durban
  - Wits Reproductive Health and HIV Institute Research Centre, Johannesburg
- Uganda (2):
  - Makerere University - Johns Hopkins University Research Collaboration Clinical Research Center, Kampala
  - MU-JHU Research Collaboration, Kampala
- Zimbabwe (3):
  - Seke South Clinical Research Center, Harare
  - Spilhaus Clinical Research Center, Harare
  - Zengeza Clinical Research Center, Harare

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baeten JM, Palanee-Phillips T, Mgodi NM, Mayo AJ, Szydlo DW, Ramjee G, Gati Mirembe B, Mhlanga F, Hunidzarira P, Mansoor LE, Siva S, Govender V, Makanani B, Naidoo L, Singh N, Nair G, Chinula L, Parikh UM, Mellors JW, Balan IC, Ngure K, van der Straten A, Scheckter R, Garcia M, Peda M, Patterson K, Livant E, Bunge K, Singh D, Jacobson C, Jiao Y, Hendrix CW, Chirenje ZM, Nakabiito C, Taha TE, Jones J, Torjesen K, Nel A, Rosenberg Z, Soto-Torres LE, Hillier SL, Brown ER; MTN-025/HOPE Study Team. Safety, uptake, and use of a dapivirine vaginal ring for HIV-1 prevention in African women (HOPE): an open-label, extension study. Lancet HIV. 2021 Feb;8(2):e87-e95. doi: 10.1016/S2352-3018(20)30304-0. PMID 33539762
- [Derived] Kutner BA, Giguere R, Lentz C, Kajura-Manyindo C, Dolezal C, Butheliezi S, Gwande M, Nampiira S, Ndlovu T, Mvinjelwa P, Mwenda W, Balan IC. Sharing Objective Measures of Adherence to a Vaginal Microbicide Promotes Candor About Actual Use and Bolsters Motivation to Prevent HIV. AIDS Behav. 2021 Mar;25(3):721-731. doi: 10.1007/s10461-020-03026-6. Epub 2020 Sep 12. PMID 32920652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: MTN-025 was implemented as a follow-on trial to MTN-020, and the inclusion and exclusion criteria were used to ensure the appropriate selection of trial participants for MTN-025.
  The Decliner Population were former MTN-020 participants who declined participation in the main MTN-025 trial, and who met the inclusion and exclusion criteria Women in the Decliner Population were invited to complete a single visit which consisted of behavioral assessments.
Pre-assignment Details: Participants were recruited from RC cohorts of MTN-020 participants. Efforts were made by RCs to maintain contact with MTN-020 (ASPIRE) participants between the end of follow-up in MTN-020 and the initiation of the MTN-025 trial (HOPE) to provide MTN-020 trial results and information regarding the HOPE trial to participants.
Groups:
- HIV Open-label Prevention: Following demonstration of safety and efficacy of the dapivirine vaginal ring in MTN-020, eligible MTN-020 participants will be offered enrollment into MTN-025, a trial designed to obtain additional safety and adherence data in women
  MTN-020: NCT01617096 MTN-025: NCT02858037
  Dapivirine Vaginal Ring: Dapivirine Vaginal Ring, 25 ring given monthly for at least one year.
Period: Overall Study
Arm/Group | HIV Open-label Prevention
Started | 1456
Exposed Primary Cohort | 1368
Completed | 1404
Not Completed | 52
Not completed — Death | 1
Not completed — Withdrawal by Subject | 18
Not completed — Participant Relocated, no follow-up planned | 26
Not completed — Lost to Follow-up | 3
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Groups:
- HIV Open-label Prevention: Following demonstration of safety and efficacy of the dapivirine vaginal ring in MTN-020, eligible MTN-020 participants will be offered enrollment into MTN-025, a trial designed to obtain additional safety and adherence data in women
  MTN-020:NCT01617096 MTN-025: NCT02858037
  Dapivirine Vaginal Ring: Dapivirine Vaginal Ring, 25 ring given monthly for at least one year.
Arm/Group | HIV Open-label Prevention
Number analyzed (Participants) | 1456
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.0 (6.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1456
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1276
  White | 0
  More than one race | 88
  Unknown or Not Reported | 84
Region of Enrollment [Number; unit: participants]
  Malawi | 157
  South Africa | 705
  Uganda | 172
  Zimbabwe | 422
Marital Status [Count of Participants; unit: Participants]
  Not Married | 770
  Married | 686

OUTCOME MEASURES:

1. Primary Outcome: The Safety Profile Associated With the Open-label Use of the Dapivirine Vaginal Matrix Ring (25 mg) in Women
Description: Number of participants Grade 2, Grade 3, and all serious Adverse Events.
Time Frame: 13 months
Population: Exposed Primary Cohort - included all participants enrolled in the Main Trial Population
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Open-label Prevention
Number analyzed (Participants) | 1368
Participants
  At least one Grade 3 or higher AE | 52
  At least one serious AE | 19
  At least one grade 2 or higher related AE | 2

2. Primary Outcome: Adherence to the Open Label Use of the Dapivirine Vaginal Matrix Ring (25 mg) in Women
Description: By measuring the residual levels of dapivirine in returned used vaginal rings.
Time Frame: 13 months
Population: Exposed Human Immunodeficiency Virus Incidence and Adherence Cohort
Measure: Mean (Full Range); unit: mg
Arm/Group | HIV Open-label Prevention
Number analyzed (Participants) | 1365
mg
  Enrollment | 21.0 [17.7 to 25.9]
  Month 1 | 21.1 [17.0 to 26.3]
  Month 2 | 21.0 [16.5 to 27.1]
  Month 3 | 21.1 [16.4 to 27.8]
  Month 6 | 21.2 [16.6 to 27.3]
  Month 9 | 21.3 [15.8 to 27.1]

3. Secondary Outcome: Incidence of HIV-1 Infection
Description: HIV-1 infection as measured by the protocol algorithm
Time Frame: 13 months
Population: Exposed Human Immunodeficiency Virus Incidence and Adherence Cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | HIV Open-label Prevention
Number analyzed (Participants) | 1365
events per 100 person-years | 2.7

4. Secondary Outcome: Number of Participant Who Acquired HIV-1 With HIV-1 Drug Resistance Associated Mutations.
Description: HIV-1 drug resistance mutations among participants who acquire HIV-1, as measured by standard genotype analysis and more sensitive methods to detect low frequency drug-resistant variants
Time Frame: 13 months
Population: Virology Population - included all HIV-1 infected participants in the Exposed HIV Incidence and Adherence Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Open-label Prevention
Number analyzed (Participants) | 33
Participants | 6

ADVERSE EVENTS:
Time Frame: 13 months
Description: Treatment-emergent Adverse Events in ≥ 2.0% of Overall Participants by System Organ Class and Preferred Term, Regardless of Severity and Causality - Exposed Primary Cohort
Arm/Group | HIV Open-label Prevention
All-Cause Mortality (participants affected / at risk) | 1/1368
Serious Adverse Events (participants affected / at risk) | 19/1368
Other Adverse Events (participants affected / at risk) | 844/1368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Open-label Prevention (N=1368)
Gastrtitis (Gastrointestinal disorders) | 1
Pelvic Inflammatory Disease (Infections and infestations) | 1
Pneummonia (Infections and infestations) | 1
Respiratory Track Infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1
Psychotic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Open-label Prevention (N=1368)
Bacteria vaginosis (Infections and infestations) | 70
Genitourinary chlamydia infection (Infections and infestations) | 115
Genitourinary tract gonococcal infection (Infections and infestations) | 58
Malaria (Infections and infestations) | 28
Upper respiratory tract infection (Infections and infestations) | 67
Urinary Tract Infection (Infections and infestations) | 71
Vulvovaginal Candidiasis (Infections and infestations) | 65
Vulvovaginitis trichomonal (Infections and infestations) | 81
ALT increased (Investigations) | 34
AST increased (Investigations) | 28
Metrorrhagia (Reproductive system and breast disorders) | 36
Pelvic pain (Reproductive system and breast disorders) | 45
Vaginal discharge (Reproductive system and breast disorders) | 110
Vulvovaginal pruritus (Reproductive system and breast disorders) | 54

LIMITATIONS AND CAVEATS:
Interpretation of the HIV-1 incidence rates is limited by the lack of a concurrent placebo group in MTN-025.

Dapivirine residual levels in returned used rings do not provide adherence information at the time of potential exposure to and infection with HIV, eg, if a participant temporarily removes the DVR during sexual intercourse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02858037/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02858037/SAP_001.pdf